CLINICAL TRIAL: NCT02596698
Title: Mitochondrial Dysfunction, Inflammation, and White Matter Integrity in Youth With Mood Disorders
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Ontario Mental Health Foundation (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1507M75201
Record Dates: First submitted 2015-10-13; First posted 2015-11-04 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Depression; Bipolar Disorder; Bipolar Disorder Not Otherwise Specified; Unspecified Mood Disorder
Keywords: Mood Disorder
MeSH Terms: conditions — Depression; Bipolar Disorder; Mood Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will keep de-identified saliva and blood samples for analysis until the completion of the study. Samples will then be destroyed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adolescents with Mood Disorders: Teens aged 13-18 with a diagnosis of a mood disorder.
- Adolescents with no Mental Health Diagnoses: 13-18, no psychiatric d/o diagnosis

SUMMARY:
This study consists of three separate appointments including a clinical assessment (interview and questionnaires), a blood draw, a social stress test, and a brain MRI.

DETAILED DESCRIPTION:
This is a research study looking at the biology of mood disorders in youth. The investigator ask participants to come in for three visits. The first visit includes a diagnostic interview, some questionnaires, and a blood draw. The blood draw will take place at the Fairview Outpatient Lab. A trained technician will take about 4 teaspoons of blood from the participant's arm. This sample will be sent to Dr. Andreazza in Toronto, Ontario for further analysis. No results will be shared with the participant.

The second visit would take place at the Fairview Riverside Ambulatory Research Center (ARC). This appointment will include the Trier Social Stress Test (TSST). For this, participants will be asked to prepare a short speech for 5 minutes and deliver that speech for in front of an audience with another task to follow. This task will be videotaped. After the participant has completed the speech task, the participant will be asked to complete a number of laptop games which will test for things like attention and memory. Participants will be asked to provide 5 saliva samples throughout the course of this visit so the investigators can look at Cortisol which is a hormone naturally found in saliva. The investigators will also ask participants to complete an additional set of 5 spit samples at home during the course of a normal day and bring those back to their next appointment.

The third visit would take place at the Center for Magnetic Resonance Research (CMRR) and would include a brain MRI. The MRI scan is noninvasive and takes about 2 hours. Participants will be asked to provide a urine sample and complete a urine toxicology screen (drug test) and pregnancy test (if female) prior to the MRI scan. Participants may not participate if drug or pregnancy testing is positive. The MRI involves taking pictures of the brain, from which measures of the integrity of certain brain tissues can be derived. For the scan, participants will be asked to lie down quietly on a scanner bed. Once they are inside the scanner, it will start to take pictures. While in the scanner, participants will be doing things like resting, or listening to music.

ELIGIBILITY:
Inclusion Criteria - All Participants:

* Age 13-18 years old
* Both child and guardian are English speaking

Inclusion Criteria - Patient Group:

* Has a diagnosis of a depressive disorder, a bipolar spectrum disorder (type 1, type 2, Unspecified), or an unspecified mood disorder based on the Diagnostic Statsitical Manual 5 (DSM-5)

Inclusion Criteria - Healthy Controls

* Does not meet criteria for any psychiatric disorders based on the DSM-5
* Does not have a family history of psychotic or mood disorders in first degree relative

Exclusion Criteria:

* Past history of brain damage, a seizure disorder, increased intracranial pressure, history of head trauma with loss of consciousness for >15 minutes, history of stroke, mental retardation, or other serious neurological disorder
* MRI contraindications such as braces, metal implants, implanted medical devices, or claustrophobia
* Intelligence quotient < 80
* Severe or acute medical illness
* A history of current (past 3 months) substance disorder (defined by DSM-5) with the exception of Nicotine
* Refusal to cooperate with study procedures
* Active suicidal ideation with intent
* Self-injury that requires medical attention (e.g. stitches) or gets significantly worse during the course of the study

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents with mood disorders will be recruited from the University of Minnesota outpatient and inpatient clinical services, through physician referral, and through community postings. Recruitment of healthy controls will be done through flyers and online postings in the community.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2015-10-31 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Blood Analysis | Baseline
  Blood samples will be analysed for mitochondrial dysfunction and resulting oxidative damage to lipids, and protein and messenger ribonucleic acid levels of inflammatory cytokines

SECONDARY OUTCOMES:
MRI Data | Up to 6 weeks after baseline
  White matter integrity. Diffusion imaging data will be processed, following registration and motion correction, using a probabilistic tractography approach that will define and extract parameters such as fractional anisotrophy and radial diffusion from fiber bundles of interest. In this study we will focus on white matter tracts connecting fronto-limbic brain regions. Details about the tractography procedures can be found at http://surfer.nmr.mgh.harvard.edu/fswiki/Tracula
Saliva Cortisol | Up to 6 weeks of baseline
  Stress Functioning. Saliva samples from the Trier Social Stress Test will be stored in a freezer and sent as a complete batch to Trier, Germany. We will conduct repeated measures ANOVA tests on the cortisol data and examine group and group x time interactions. We will calculate the Area Under the Curve for each person's pattern of cortisol responses over time, and these values will be used in multivariate regression analyses below.
Beck Depression Inventory (BDI-II) | Baseline and within 6 weeks of baseline
  Measures levels of depression in participants. Has information on suicidal ideation. If participants are suicidal, a member of research staff will talk with the participant and develop a safety plan with the adolescent and their parent.
Children's Depression Rating Scale - Revised (CDRS-R) | Baseline
  Measures levels of depression in participants. Has information on suicidal ideation. If participants are suicidal, a member of research staff will talk with the participant and develop a safety plan with the adolescent and their parent.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn R Cullen, MD, Principal Investigator — University of Minnesota; Ana Andreazza, PhD, Principal Investigator — University of Toronto, Ontario; Bonnie Klimes-Dougan, PhD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Ambulatory Research Center (ARC), Minneapolis, Minnesota
  - Center for Magnetic Resonance Research, Minneapolis, Minnesota